CLINICAL TRIAL: NCT01080131
Title: A Randomized, Controlled Study of ACZ885 (Canakinumab) on the Treatment and Prevention of Gout Flares in Patients With Frequent Flares for Whom NSAIDs and/or Colchicine Are Contraindicated, Not Tolerated or Ineffective Including a 12 Weeks Extension Study and a 1 Year Open-label Extension Study
Brief Title: Canakinumab in the Treatment of Acute Gout Flares and Prevention of New Flares in Patients Unable to Use Non-steroidal Anti-inflammatory Drugs (NSAIDs) and/or Colchicines Including a 12 Week Extension and a 1 Year Open-label Extension Study.
Acronym: β-RELIEVED-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885H2357; 2010-018913-32 (EudraCT Number); CACZ885H2357E1 (Other: Novartis); NCT01137344 (obsolete NCT alias); NCT01194921 (obsolete NCT alias)
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2011-12-26 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-04

CONDITIONS: Acute Gout
Keywords: Frequent flares; Gout; Anti-interleukin-1β monoclonal antibody
MeSH Terms: conditions — Gout | interventions — canakinumab; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Canakinumab 150 mg (Experimental): Participants received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Participants could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Participants completing the 12 week core study could continue to be treated in a 12 week extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  In the second extension study participants were to receive open-label on demand treatment with canakinumab 150 mg sc upon new flare for 1 year, for a total duration of 18 months.
  Interventions: Drug: Canakinumab 150 mg; Drug: Placebo to triamcinolone acetonide
- Triamcinolone acetonide 40 mg (Active Comparator): Participants received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 subcutaneous (sc) injection of placebo to canakinumab on Day 1. Participants could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Participants completing the 12 week core study could continue to be treated in a 12 week extension study for any new gout flare on demand with the same treatment as assigned in the core study.
  In the second extension study participants were to switch to open-label on demand treatment with canakinumab 150 mg sc upon new flare for 1 year. Triamcinolone acetonide was not to be administered in the second extension study.
  Interventions: Drug: Triamcinolone acetonide 40 mg; Drug: Placebo to canakinumab

INTERVENTIONS:
Drug: Canakinumab 150 mg — Canakinumab 150 mg was supplied in 6 mL glass vials each containing nominally 150 mg canakinumab (plus 20% overfill).
  Arms: Canakinumab 150 mg
Drug: Triamcinolone acetonide 40 mg — Triamcinolone acetonide 40 mg was supplied as a suspension.
  Arms: Triamcinolone acetonide 40 mg
Drug: Placebo to canakinumab — Placebo to canakinumab was supplied in 6 mL glass vials containing placebo powder as a lyophilized cake.
  Arms: Triamcinolone acetonide 40 mg
Drug: Placebo to triamcinolone acetonide — Placebo triamcinolone acetonide was supplied as a lipid emulsion similar in appearance to triamcinolone acetonide.
  Arms: Canakinumab 150 mg

SUMMARY:
The purpose of this study was to demonstrate that canakinumab given upon acute gout flares relieves the signs and symptoms and prevents recurrence of gout flares in patients with frequent flares of gout for whom non-steroidal anti-inflammatory drugs (NSAIDs) and/ or colchicine are contraindicated, not tolerated, or ineffective. The efficacy of canakinumab was compared to the corticosteroid triamcinolone acetonide.

The purpose of the first 12 week extension study was to collect additional safety, tolerability and efficacy data in patients who have completed the core study CACZ885H2357.

The purpose of the second one year open-label extension study was to confirm the long-term safety and tolerability of canakinumab in patients who had completed the first extension study.

ELIGIBILITY:
Core Study:

Inclusion criteria:

* Meeting the American College of Rheumatology (ACR) 1977 preliminary criteria for the classification of acute arthritis of primary gout
* Onset of current acute gout flare within 5 days prior to study entry
* Baseline pain intensity ≥ 50 mm on the 0-100 mm visual analog scale (VAS)
* History of ≥ 3 gout flares within the 12 months prior to study entry
* Contraindication, or intolerance, or lack of efficacy for non-steroidal anti-inflammatory drugs (NSAID) and/or colchicine

Exclusion criteria:

* Rheumatoid arthritis, evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis
* Presence of severe renal function impairment
* Use of specified pain relief medications or biologics (corticosteroids, narcotics, paracetamol/acetominophen, ibuprofen, colchicine, IL-blocker, and tumor necrosis factor inhibitor within specified periods prior to study entry
* Live vaccinations within 3 months prior to randomization
* Requirement for administration of antibiotics against latent tuberculosis (TB)
* Refractory heart failure (Stage D)
* Unstable cardiac arrhythmias or unstable symptomatic coronary ischemia
* Any active or recurrent bacterial, fungal, or viral infection

Extension Study 1:

Inclusion:

- Completion of the Core study. A patient was defined as completing the core study if they completed the study up to and including visit 7.

Exclusion:

- Continuation in this extension study was considered inappropriate by the treating physician.

Extension Study 2:

Inclusion Criteria:

* Completion of the first extension study CACZ885H2357E1. A patient was defined as completing the first extension study if they completed the study up to and including Visit 10).

Exclusion Criteria:

-Continuation in this second extension study was considered inappropriate by the treating physician.

Other protocol-defined inclusion-exclusion criteria applied to the core and extension studies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (107):
- United States (95):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Novartis Investigative site, Foley, Alabama
  - Horizon Research Group, Inc., Mobile, Alabama
  - Sun Valley Arthritis Center, Ltd, Peoria, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - Providence Research, Burbank, California
  - Diagnamics, Inc., Carlsbad, California
  - Med Investigations, Fair Oaks, California
  - Valerius Medical Group and Research Center of Long Branch, Long Beach, California
  - Lucita M. Cruz, M.D., Inc., Norwalk, California
  - Sierra Clinical Research, Orangevale, California
  - Chaparral Medical Grp, INC Clinical Research, Pomona, California
  - River City Clinical Research, Sacramento, California
  - Arthritis Associates, San Antonio, California
  - California Research Foundation, San Diego, California
  - Rochester clinical Research, San Diego, California
  - Ritchken and First MDs, San Diego, California
  - Huntington Medical Foundation, San Marino, California
  - Crest Clinical Trials, Santa Ana, California
  - Orange County Research Center, Tustin, California
  - Progressive Clinical Research, Vista, California
  - Center for Clinical Trials of San Gabriel, West Covina, California
  - Clinical Res Ct of CT - Arthritis Associates of CT/NY, LLC, Danbury, Connecticut
  - Innovative Research of West Florida, Clearwater, Florida
  - Health Awareness, Jupiter, Florida
  - Pines Research, LLC Pembroke Clinical Trials, Pembroke Pines, Florida
  - DMI Healthcare Group, Inc., Pinellas Park, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - RST DAta Research, Conyers, Georgia
  - Q Clinical Research, Decatur, Georgia
  - Harbin Clinic, Rome, Georgia
  - Sonora Clinical Research, LLC, Boise, Idaho
  - Northwest Clinical Trials, Boise, Idaho
  - The Arthritis Center, Springfield, Illinois
  - Deaconess Clinic, Evansville, Indiana
  - Pinnacle Medical Research, Overland Park, Kansas
  - Wichita Clinic, Wichita, Kansas
  - Dolby Research, LLC, Baton Rouge, Louisiana
  - Gulf Coast Research, LLC, Lafayette, Louisiana
  - Clinical Trials Management, Metairie, Louisiana
  - Arthritis and Diabetes Clinic, Monroe, Louisiana
  - Regional Research Specialists, Shreveport, Louisiana
  - The Family Doctors, Shreveport, Louisiana
  - Center for Rheumatology & Bone Research, Wheaton, Maryland
  - MASS Research, LLC, Waltham, Massachusetts
  - Clarkston Medical Group, Clarkston, Michigan
  - L Kage Healthcare Services, Flint, Michigan
  - West Michigan Rheumatology, Grand Rapids, Michigan
  - *Private Practice*, Lansing, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Arthritis Associates of Mississippi, Jackson, Mississippi
  - CRC of Jackson, Jackson, Mississippi
  - Phillips Medical Center, Jackson, Mississippi
  - Montana Medical Research, Missoula, Montana
  - Quality Clinical Research, Omaha, Nebraska
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - Clinical Research Advantage, Inc, Henderson, Nevada
  - Arthritis and Osteoporosis Associates, Freehold, New Jersey
  - UMDNJ Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Arthritis and Osteoporosis Medical Association, Brooklyn, New York
  - Andrew J. Porges, MD, PC, Roslyn, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - The Center For Nutrition and Preventive Medicine, Charlotte, North Carolina
  - Unifour Medical Research Associates, Hickory, North Carolina
  - Jones Family Practice, PA, Shelby, North Carolina
  - Columbia Arthritis Center, Columbus, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - Ohio Clinical Research, LLC, Willoughby Hills, Ohio
  - Humility of Mary Health Partners DBA St. Elizabeth Health Ce, Youngstown, Ohio
  - Health Research of Oklahoma, PLLC, Oklahoma City, Oklahoma
  - Health Research Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Philadelphia VA medical Center, Philadelphia, Pennsylvania
  - Partners in Clinical Research, Bumberland, Rhode Island
  - Medical Research South, Charleston, South Carolina
  - Pharmacorp Clinical Trials, INC, Charleston, South Carolina
  - Tlm Medical Services Llc, Columbia, South Carolina
  - Palmetto Clinical Trial Services, LLC, Greenville, South Carolina
  - Community Research Partners, Inc., Varnville, South Carolina
  - Tri-Cities Medical Research, Bristol, Tennessee
  - Alpha Clinical Research, Clarksville, Tennessee
  - The Jackson Clinic, Jackson, Tennessee
  - The Arthritis Clinic, Jackson, Tennessee
  - MultiSpecialty Clinical Research, Johnson City, Tennessee
  - Lovelace Scientific Resource, Austin, Texas
  - Rheumatic Disease Clinical Research Center, Llc, Houston, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Leander Healthcare Center, Leander, Texas
  - Accurate Clinical Research, Nassau Bay, Texas
  - North Hills Family Practice, North Richard Hills, Texas
  - Arthritis Center South Texas, San Antonio, Texas
  - Novartis Investigative site, Danville, Virginia
  - Health Research of Hampton Roads, Newport News, Virginia
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative site, Sainte-Foy, Quebec
- China (4):
  - Novartis Investigative Site, Kaohsiung Hsien, Taiwan
  - Novartis Investigative Site, Kaohsiung, Taiwan
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
- Netherlands (2):
  - Novartis Investigative Site, Enschede
  - Novartis Investigative site, Leeuwarden
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg

REFERENCES:
- [Derived] Chakraborty A, Van LM, Skerjanec A, Floch D, Klein UR, Krammer G, Sunkara G, Howard D. Pharmacokinetic and pharmacodynamic properties of canakinumab in patients with gouty arthritis. J Clin Pharmacol. 2013 Dec;53(12):1240-51. doi: 10.1002/jcph.162. Epub 2013 Sep 30. PMID 24122883

RESULTS

PARTICIPANT FLOW:
Groups:
- Canakinumab 150 mg: Participants received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Participants could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. In the first extension study participants completing the 12 week core study could continue to be treated on demand with the same treatment for another 12 weeks for any new gout flare.
  In the second extension study participants were to receive open-label on demand treatment with canakinumab 150 mg sc for any new flare for an additional year, for a total duration of 18 months.
- Triamcinolone Acetonide 40 mg: Participants received 1 intramuscular injection of triamcinolone acetonide 40 mg and 1 sc injection of placebo to canakinumab on Day 1. Participants could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose.
  In the first extension study participants completing the 12 week core study could continue to be treated on demand with the same treatment for another 12 weeks for any new gout flare.
  In the second extension study participants were to switch to open-label on demand treatment with canakinumab 150 mg sc for any new flare for an additional year. Triamcinolone acetonide was not to be administered in the second extension study.
Period: Core Study (0- 12 Weeks)
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Started | 112 | 114
Completed | 99 | 103
Not Completed | 13 | 11
Not completed — Abnormal laboratory value(s) | 1 | 1
Not completed — Patient withdrew consent | 6 | 4
Not completed — Lost to Follow-up | 5 | 3
Not completed — Administrative problems | 0 | 1
Not completed — Death | 1 | 0
Not completed — Protocol deviation | 0 | 2
Period: Extension Study 1 (12 -24 Weeks)
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Started | 84 | 76
Completed | 78 | 72
Not Completed | 6 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Unsatisfactory Therapeutic Effect | 0 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 1 | 0
Period: Extension Study 2 (25-72 Weeks)
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Started | 72 | 65
Re-treated With or Switch to Canakinumab | 62 (Includes patients re-treated with canakinumab at any time during the 72 weeks) | 41 (Includes patients switched to canakinumab from Week 25 - Week 72)
Completed | 64 | 54
Not Completed | 8 | 11
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg | Total
Number analyzed (Participants) | 112 | 114 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (12.10) | 52.6 (12.28) | 51.6 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 100 | 105 | 205

OUTCOME MEASURES:

1. Primary Outcome: Time to First New Flare: Survival Analysis During the 12 Weeks of Study
Description: Kaplan-Meier estimates of time to first new flare and confidence intervals were determined. For patients with event, time to event = (date of event - date of first dose of study drug + 1). Patients met definition of new flare if they had: •Flare in joint, not a previously affected joint (at baseline or during study) •Flare in joint previously affected (at baseline or during study) after previous flare in joint has resolved completely. Patients did not meet criterion of having new gout flare if: • Increasing/renewed gout pain in an affected joint before flare has resolved completely.
Time Frame: Baseline to 12 weeks
Population: Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Canakinumab 150 mg: Participants received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Participants could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose.
- Triamcinolone Acetonide 40 mg: Participants received 1 intramuscular injection of triamcinolone acetonide 40 mg and 1 sc injection of placebo to canakinumab on Day 1. Participants could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose.
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
Days | NA [NA to NA] — A median time to first new flare could not be estimated because <50% patients had a new flare during the time period. | NA [NA to NA] — A median time to first new flare could not be estimated because <50% patients had a new flare during the time period.

2. Secondary Outcome: Time to at Least a 50% Reduction in Self-assessed Pain Intensity in the Joint Most Affected at Baseline Measured on a Visual Analog Scale (VAS)
Description: Kaplan-Meier estimates of the time to at least a 50% reduction in self-assessed pain intensity in the joint most affected at Baseline and the confidence intervals were determined along with 95% confidence interval. Patients scored their pain intensity on a 0-100 mm VAS, ranging from no pain (0) to unbearable pain (100). Scores on the 100 mm linear scale were measured to the nearest millimeter from the left. Pain was scored at Baseline; at 6 and 12 hours post-dose; and at 1, 2, 3, 4, 5, 6, and 7 days post-dose.
Time Frame: Baseline to 7 days post-dose (randomization)
Population: Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. Last Observation Carried Forward (LOCF) method was used to impute post dose measurement.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 111 | 109
hours | 25.0 [23.0 to 48.0] | 48.0 [24.0 to 49.0]

3. Secondary Outcome: Time to Complete Resolution of Pain; Survival Analysis
Description: Kaplan-Meier estimates of the time to complete resolution of self-assessed pain intensity in the joint most affected and the confidence interval was determined. Patients scored their pain intensity on a 5-point Likert scale (none, mild, moderate, severe, extreme). Pain was scored at Baseline; 6 and 12 hours; 1, 2, 3, 4, 5, 6, and 7 days post-dose.
Time Frame: Baseline to 7 days post-dose (randomization)
Population: Full Analysis Set (FAS): All patients that received study drug.
Measure: Number (95% Confidence Interval); unit: hours
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
hours | 144.0 [120 to NA] — The upper limit was not estimable in the study as it is longer than duration of study. | NA [168 to NA] — The median time to complete resolution could not be estimated because <50% of patients had a complete resolution during the time period.

4. Secondary Outcome: SF 36 Physical Function Score at Week 12
Description: SF-36 measures impact of disease on overall quality of life (QoL). 36-item survey has 8 subscales that can be aggregated into physical and mental component summary scores. Scores are standardized with the use of norm-based methods based on assessment of the general U.S. population free of chronic conditions. Scores range from 1-100 with a mean=50 and a standard deviation=10. A higher score indicates less impact on QoL. Analysis of covariance (ANCOVA) model was used with treatment group and baseline SF-36 physical function subscore as covariates.
Time Frame: Week 12
Population: Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. Participants with observations at Week 12 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 83 | 81
Units on a scale | 81.46 (2.786) | 78.75 (2.820)

5. Secondary Outcome: Percentage of Participants With at Least 1 New Gout Flare During the 12 Weeks of the Study
Description: The percentage of participants who experienced at least 1 new gout flare during the 12 week study treatment period.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
percentage of participants | 13.4 | 36.8

6. Primary Outcome: Self-assessed Pain Intensity in the Joint Most Affected at Baseline Measured on a Visual Analog Scale (VAS) at 72 Hours Post-dose
Description: Patients scored their pain intensity in the joint most affected at Baseline on a 0-100 mm VAS, ranging from no pain (0) to unbearable pain (100), at 72 hours post-dose. Scores on the 100 mm linear scale were measured to the nearest millimeter from the left. The analysis of covariance (ANCOVA) analysis included treatment group, Baseline VAS score, and body mass index (BMI) at Baseline as covariates.
Time Frame: 72 hours post-dose (randomization)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 111 | 109
mm | 22.1 (2.33) | 31.9 (2.35)

7. Secondary Outcome: Pharmacokinetic Concentrations
Description: Canakinumab concentration was analyzed in serum by means of a competitive Enzyme-linked immunosorbent assay (ELISA) assay with a lower limit of quantification (LOQ) at 100 ng/mL.
Time Frame: 12 weeks post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Canakinumab 150 mg: Patients received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Patients could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. Patients completing the 12 weeks core study were allowed to continue to be treated in another 12 weeks extension study for any new gout flare on demand with the same treatment as assigned in the core study.
Arm/Group | Canakinumab 150 mg
Number analyzed (Participants) | 99
µg/mL | 2.16 (2.375)

8. Secondary Outcome: Self-assessed Pain Intensity in the Joint Most Affected at Baseline Measured on a Visual Analog Scale (0-100 mm VAS)
Description: Patients scored their pain intensity in the joint most affected at Baseline on a 0-100 mm VAS, ranging from no pain (0) to unbearable pain (100), from 6 hours to 7 days post-dose. Scores on the 100 mm linear scale were measured to the nearest millimeter from the left. The ANCOVA analysis included treatment group, Baseline VAS score, and body mass index (BMI) at Baseline as covariates.
Time Frame: 6, 12, 24, 48, and 72 hours; and 4, 5, 6, and 7 days post-dose (randomization)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
mm
  6 hours post-dose | 58.7 (1.94) | 60.3 (1.96)
  12 hours post-dose | 50.8 (2.16) | 52.0 (2.18)
  24 hours post-dose | 39.1 (2.39) | 45.0 (2.41)
  48 hours post-dose | 29.5 (2.45) | 38.9 (2.48)
  72 hours post-dose | 22.1 (2.33) | 31.9 (2.35)
  4 days post-dose | 19.2 (2.25) | 27.7 (2.27)
  5 days post-dose | 16.4 (2.23) | 25.4 (2.25)
  6 days post-dose | 14.3 (2.20) | 22.3 (2.22)
  7 days post-dose | 14.0 (2.18) | 19.5 (2.20)

9. Secondary Outcome: Self-assessed Pain Intensity in the Joint Most Affected at Last Post-Baseline Measured on a Visual Analog Scale (VAS)
Description: Patient's assessment of gout pain intensity in the most affected joint (on a 0-100 mm VAS) for the last post-baseline flare, ranging from no pain (0) to unbearable pain (100), was summarized up to 7 days after receiving a re-dose of study drug by time point. Scores on the 100 mm linear scale were measured to the nearest millimeter from the left. The covariance analysis included treatment group, Baseline VAS score at that flare, and body mass index (BMI) at Baseline as covariates.
Time Frame: 6, 12, 24, 48, and 72 hours; and 4, 5, 6, and 7 days post-dose for last post-baseline flare that occurred up until the end of the first extension study (24 weeks).
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. For assessments made up to 7 days after re-dosing, pain values were imputed using the Last- Observation-Carried-Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: mm
Groups:
- Canakinumab 150 mg: Participants received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Participants could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. In the first extension study participants completing the 12 week core study could continue to be treated on demand with the same treatment for another 12 weeks for any new gout flare.
- Triamcinolone Acetonide 40 mg: Participants received 1 intramuscular injection of triamcinolone acetonide 40 mg and 1 sc injection of placebo to canakinumab on Day 1. Participants could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose.
  In the first extension study participants completing the 12 week core study could continue to be treated on demand with the same treatment for another 12 weeks for any new gout flare.
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 25 | 46
mm
  6 hours post-dose | 57.4 (3.07) | 59.1 (2.26)
  12 hours post-dose | 50.7 (4.24) | 53.3 (3.12)
  24 hours post-dose | 46.2 (4.74) | 43.8 (3.49)
  48 hours post-dose | 42.3 (4.96) | 34.2 (3.65)
  72 hours post-dose | 37.0 (5.12) | 26.1 (3.77)
  4 days post-dose | 31.3 (4.75) | 23.4 (3.49)
  5 days post-dose | 29.0 (5.11) | 21.6 (3.76)
  6 days post-dose | 28.1 (5.04) | 20.5 (3.71)
  7 days post-dose | 24.1 (5.03) | 19.1 (3.70)

10. Secondary Outcome: Time to the First New Gout Flare During 24 Weeks
Description: Kaplan-Meier (KM) estimates of the time to first new flare and confidence intervals were determined. Participants met the definition of a new flare if they had:
  * Flare in joint, not a previously affected joint (at baseline or during study)
  * Flare in joint previously affected (at baseline or during study) after previous flare in joint has resolved completely.
  Participants did not meet the criterion of having a new gout flare if they had increasing/renewed gout pain in an affected joint before the flare had resolved completely.
Time Frame: From randomization to the end of the first extension period (24 weeks).
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
days | NA [NA to NA] — Not estimable due to the low number of events at the time of the assessment (24 weeks). | 146 [94.0 to NA] — Not estimable due to the low number of events at the time of the assessment (24 weeks).

11. Secondary Outcome: Mean Number of New Gout Flares Per Patient During 24 Weeks
Description: Patients met definition of new flare if they had:
  * Flare in joint, not a previously affected joint(at baseline or during study)
  * Flare in joint previously affected (at baseline or during study) after previous flare in joint has resolved completely.
  Participants did not meet the criterion of having a new gout flare if they had increasing/renewed gout pain in an affected joint before the flare had resolved completely.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: new flares per patient
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
new flares per patient | 0.35 (0.694) | 0.80 (1.115)

12. Secondary Outcome: Time to First Intake of Rescue Medication
Description: Participants who had difficulty in tolerating their pain were allowed to take rescue medication after the 6-hour post-dose pain assessments as follows:
  * Acetaminophen (paracetamol) 500 mg and/ or codeine 30 mg as required. A maximum of 1 g/dose or 3 g/day of acetaminophen and 30 mg/ dose or 180 mg/day of codeine was allowed.
  * If they had insufficient pain relief, participants were allowed to take a maximum of 30 mg of oral prednisolone as required per day for 2 days followed by up to 20 mg of prednisolone as required subsequent days within 7 days of a gout flare.
  Use of these treatments during the first 7 days of a gout flare was recorded as rescue medication.
  Kaplan-Meier estimates of the time to first intake of rescue medication, in hours, and the confidence interval were determined for the flare experienced at study entry (Baseline flare) and the last new flare (last post-baseline flare) that occurred up until the end of the first extension period (24 weeks).
Time Frame: For 7 days after the first dose for the baseline flare and 7 days post-dose for the last post-baseline flare that occurred up until the end of the first extension study (24 weeks).
Population: For the Baseline flare the population analyzed consisted of the Full Analysis Set (FAS). For the last post-baseline flare the population analyzed consisted of patients re-treated for at least one new flare. Patients who did not take rescue medication had the time-to-first rescue medication intake censored at 7 days post dosing and re-dosing.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
hours
  Baseline flare [N= 112, 114] | NA [24 to NA] — The data were not estimable as <50% patients took rescue medication | 37.5 [14 to NA] — Upper bound did not cross the median value hence the upper limit was not estimable.
  Last post-baseline flare [N=25, 46] | 32 [8.0 to NA] — Upper bound did not cross the median value hence the upper limit was not estimable. | NA [12.0 to NA] — The data were not estimable as <50% patients took rescue medication

13. Secondary Outcome: Percentage of Participants Who Took Rescue Medication
Description: Participants who had difficulty in tolerating their pain were allowed to take rescue medication after the 6-hour post-dose pain assessments as follows:
  * Acetaminophen (paracetamol) 500 mg and/ or codeine 30 mg as required. A maximum of 1 g/dose or 3 g/day of acetaminophen and 30 mg/ dose or 180 mg/day of codeine was allowed.
  * If they had insufficient pain relief, participants were allowed to take a maximum of 30 mg of oral prednisolone as required per day for 2 days followed by up to 20 mg of prednisolone as required subsequent days within 7 days of a gout flare.
  Use of these treatments during the first 7 days of a gout flare was recorded as rescue medication.
Time Frame: as for outcome 12
Population: For the Baseline flare the population analyzed consisted of the Full Analysis Set (FAS). For the last post-baseline flare the population analyzed consisted of patients re-treated for at least one new flare.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
percentage of participants
  Baseline flare [N= 112, 114] | 43.8 | 57.0
  Last post-baseline flare [N=25, 46] | 56.0 | 41.3

14. Secondary Outcome: Amount of Rescue Medication Taken
Description: Patients who had difficulty in tolerating their pain were allowed to take rescue medication after the 6-hour post-dose pain assessments as follows:
  * Acetaminophen (paracetamol) 500 mg and/ or codeine 30 mg as required. A maximum of 1 g/dose or 3 g/day of acetaminophen and 30 mg/ dose or 180 mg/day of codeine was allowed.
  * If they had insufficient pain relief, patients were allowed to take a maximum of 30 mg of oral prednisolone as required per day for 2 days followed by up to 20 mg of prednisolone as required subsequent days within 7 days of a gout flare.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
mg
  Baseline flare: Acetaminophen [N=112, 114] | 1375.0 (2726.63) | 2526.5 (3925.13)
  Baseline flare: Codeine [N=112, 114] | 27.2 (100.40) | 60.6 (144.38)
  Baseline flare: Prednisone/Predinisone [N=112,114] | 9.2 (35.32) | 19.3 (44.88)
  Last flare: Acetaminophen [N=25, 46] | 2292.0 (3462.65) | 1541.3 (3771.33)
  Last flare: Codeine [N= 25, 46] | 64.8 (224.11) | 65.2 (178.70)
  Last flare: Prednisolone/Predinisone [N= 25, 46] | 5.6 (14.46) | 18.3 (48.00)

15. Secondary Outcome: Physician's Global Assessment of Response to Treatment
Description: The study physician made a global assessment of the patient's response to treatment using a 5-point Likert scale: Very good, good, fair, poor, very poor. The percentage of patients in each category is reported. The physician completed the assessment without viewing any of the patient's own assessments (pain intensity and patient's global assessment of response to treatment).
Time Frame: 72 hours post-dose and 24-weeks post-dose.
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. 'N' in each category indicates participants with observations available for this endpoint at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
percentage of participants
  72 hours - Very good [N= 107, 109] | 43.0 | 25.7
  72 hours - Good [N= 107, 109] | 43.0 | 35.8
  72 hours - Fair [N= 107, 109] | 11.2 | 26.6
  72 hours - Poor [N= 107, 109] | 2.8 | 6.4
  72 hours - Very poor [N= 107, 109] | 0.0 | 5.5
  24 weeks - Very good [N=79, 71] | 77.2 | 66.2
  24 weeks - Good [N=79, 71] | 16.5 | 29.6
  24 weeks - Fair [N=79, 71] | 5.1 | 4.2
  24 weeks - Poor [N=79, 71] | 1.3 | 0.0
  24 weeks - Very poor [N=79, 71] | 0.0 | 0.0

16. Primary Outcome: Number of Participants With Adverse Events, Death and Serious Adverse Events During 24 Weeks
Description: This was primary endpoint of extension study 1. Adverse event is defined as any unfavorable and unintended diagnosis, symptom sign including an abnormal laboratory finding, syndrome or disease which either occurs during the study, having been absent at baseline, or, if present at baseline, appears to worsen. A serious adverse event is defined as any untoward medical occurrence that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: During 24 weeks overall
Population: Safety population consisted of all patients who received study drug in the core study and had at least one post-baseline safety assessment
Measure: Number; unit: Participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
Participants
  Adverse event | 78 | 65
  Death | 1 | 0
  Serious adverse event | 7 | 2

17. Secondary Outcome: Patient's Global Assessment of Response to Treatment
Description: Participants made a global assessment of response to treatment using a 5-point Likert scale: Excellent, good, acceptable, slight, poor. The percentage of participants in each category is reported.
Time Frame: 72 hours post-dose and 24 weeks post-dose
Population: The Full Analysis Set (FAS) consisted of all patients as randomized in the core study who had taken at least one dose of study drug. 'N' in each category indicates participants with observations available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
percentage of participants
  72 hours - Excellent [N=108, 108] | 36.1 | 19.4
  72 hours - Good [N=108, 108] | 37.0 | 32.4
  72 hours - Acceptable [N=108, 108] | 18.5 | 13.9
  72 hours - Slight [N=108, 108] | 4.6 | 25.0
  72 hours - Poor [N=108, 108] | 3.7 | 9.3
  24 weeks - Excellent [N=79, 72] | 59.5 | 40.3
  24 weeks - Good [N=79, 72] | 26.6 | 44.4
  24 weeks - Acceptable [N=79, 72] | 6.3 | 13.9
  24 weeks - Slight [N=79, 72] | 6.3 | 1.4
  24 weeks - Poor [N=79, 72] | 1.3 | 0.0

18. Secondary Outcome: Physician's Assessment of Tenderness, Swelling, and Erythema of the Most Affected Joint
Description: The study physician assessed the most affected joint for: Tenderness on a 0-3 point scale: No pain, patient states that "there is pain", patient states "there is pain and winces", and patient states "there is pain, winces, and withdraws" on palpation or passive movement of the affected study joint; Swelling on a 0-3 point scale: No swelling, palpable, visible, and bulging beyond the joint margins; and Erythema: Present or absent. The percentage of participants in each category is reported.
Time Frame: 72 hours post-dose and 24 weeks post-dose
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
percentage of participants
  72 hours - Tenderness: No pain [N=107, 109] | 47.7 | 30.3
  72 hours - Tenderness: Pain [N=107, 109] | 43.9 | 46.8
  72 hours - Tenderness: Pain & winces [N=107, 109] | 4.7 | 14.7
  72 hours - Tenderness:Winces/withdraws [N=107,109] | 3.7 | 8.3
  24 weeks - Tenderness: No pain [N=79, 71] | 88.6 | 91.5
  24 weeks - Tenderness: Pain [N=79, 71] | 8.9 | 5.6
  24 weeks - Tenderness: Pain and winces [N=79, 71] | 1.3 | 1.4
  24 weeks - Tenderness: Winces/withdraws [N=79, 71] | 1.3 | 1.4
  72 hours - Swelling: No swelling [N=107,109] | 47.7 | 35.8
  72 hours - Swelling: Palpable [N=107,109] | 28.0 | 29.4
  72 hours - Swelling: Visible [N=107,109] | 22.4 | 28.4
  72 hours - Swelling: Bulging [N=107,109] | 1.9 | 6.4
  24 weeks - Swelling: No swelling [N=79, 71] | 93.7 | 94.4
  24 weeks - Swelling: Palpable [N=79, 71] | 5.1 | 4.2
  24 weeks - Swelling: Visible [N=79, 71] | 1.3 | 1.4
  24 weeks - Swelling: Bulging [N=79, 71] | 0.0 | 0.0
  72 hours - Erythema: Absent [N=107, 108] | 74.8 | 66.7
  72 hours - Erythema: Present [N=107, 108] | 25.2 | 33.3
  24 weeks - Erythema: Absent [N=79, 71] | 97.5 | 97.2
  24 weeks - Erythema: Present [N=79, 71] | 2.5 | 2.8

19. Secondary Outcome: Physician's Assessment of Range of Motion of the Most Affected Joint
Description: The study physician assessed the range of motion of the most affected joint for range of motion on a 5-point Likert scale: Normal, mildly restricted, moderately restricted, severely restricted, immobilized. The percentage of participants in each category is reported.
Time Frame: 72 hours post-dose and 24 weeks post-dose
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
percentage of participants
  72 hours - Normal [N=107,109] | 47.7 | 28.4
  72 hours - Mildly restricted [N=107,109] | 37.4 | 45.9
  72 hours - Moderately restricted [N=107,109] | 13.1 | 20.2
  72 hours - Severely restricted [N=107,109] | 1.9 | 5.5
  72 hours - Immobilized [N=107,109] | 0.0 | 0.0
  24 weeks - Normal [N=79, 71] | 86.1 | 97.2
  24 weeks - Mildly restricted [N=79, 71] | 10.1 | 2.8
  24 weeks - Moderately restricted [N=79, 71] | 2.5 | 0.0
  24 weeks - Severely restricted [N=79, 71] | 1.3 | 0.0
  24 weeks - Immobilized [N=79, 71] | 0.0 | 0.0

20. Primary Outcome: Number of Participants With Adverse Events, Death and Serious Adverse Events (72 Weeks Overall)
Description: This was the primary endpoint of extension study 2. An adverse event was defined as any unfavorable and unintended diagnosis, symptom sign including an abnormal laboratory finding, syndrome or disease which either occurs during the study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse event is defined as any untoward medical occurrence that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: 72 weeks
Population: as for outcome 16
Measure: Number; unit: participants
Groups:
- All Canakinumab: Participants received 1 subcutaneous (sc) injection of canakinumab 150 mg and 1 intramuscular (im) injection of placebo to triamcinolone acetonide on Day 1. Participants could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose.
  In the first extension study, participants completing the 12 week core study could continue to be treated on demand with the same study treatment for an additional 12 weeks for any new gout flare.
  In the second extension study participants were to receive open-label on demand treatment with canakinumab 150 mg sc upon new flare for 1 year, for a total duration of 18 months.
- Canakinumab: Before Retreatment: Participants who received canakinumab in the core study and were re-treated with canakinumab during the core study or extension study 1 or 2. Reported data include adverse events that occurred in this re-treated population before re-treatment with canakinumab.
- Canakinumab: After Retreatment: Participants who received canakinumab in the core study and were re-treated with canakinumab during the core study or extension study 1 or 2. Reported data include adverse events that occurred in this re-treated population after re-treatment with canakinumab.
- All Triamcinolone Acetonide: Participants received 1 intramuscular (im) injection of triamcinolone acetonide 40 mg and 1 sc injection of placebo to canakinumab on Day 1. Participants could receive a re-dose of study drug on demand upon the occurrence of new flares, but re-dosing could not occur until 14 days had elapsed after the previous dose. In the first extension study participants completing the 12 week core study could continue to be treated on demand with the same study treatment another 12 weeks for any new gout flare.
  Reported data include all adverse events that occurred during the core study and extension studies 1 and 2, before participants were switched to canakinumab.
- Triam: Before Switch to Canakinumab: Participants who were treated with triamcinolone acetonide (triam) during the core study and extension study 1 and who were switched to open-label on demand treatment with canakinumab 150 mg sc upon new flare in extension study 2. Data are reported for adverse events that occurred before the switch to canakinumab.
- Triam: After Switch to Canakinumab: Participants who were treated with triamcinolone acetonide during the core study and extension study 1 and who were switched to open-label on demand treatment with canakinumab 150 mg sc upon new flare in extension study 2. Data are reported for adverse events that occurred after the switch to canakinumab.
Arm/Group | All Canakinumab | Canakinumab: Before Retreatment | Canakinumab: After Retreatment | All Triamcinolone Acetonide | Triam: Before Switch to Canakinumab | Triam: After Switch to Canakinumab
Number analyzed (Participants) | 112 | 62 | 62 | 114 | 41 | 41
participants
  Any adverse event | 85 | 44 | 39 | 70 | 29 | 27
  Death | 1 | 0 | 0 | 0 | 0 | 0
  Serious adverse event | 12 | 1 | 5 | 4 | 0 | 3

21. Secondary Outcome: High-sensitivity C-reactive Protein (hsCRP) and Serum Amyloid A Protein (SAA) Levels
Description: High sensitivity C-reactive protein (hsCRP) and serum amyloid A (SAA) were determined in blood serum in order to identify the presence of inflammation, to determine its severity, and to monitor the response to treatment. Analyses were measured by a central laboratory. The analysis included treatment group, log-transformed protein level at baseline, and body mass index (BMI) at baseline as covariates.
Time Frame: 72 hours after the first dose for the baseline flare and 72 hours post-dose for the last post-baseline flare that occurred up until the end of the first extension study (24 weeks).
Population: For the Baseline flare the population analyzed consisted of the Full Analysis Set (FAS). For the last post-baseline flare the population analyzed consisted of patients re-treated for at least one new flare. "N" indicates the number of participants with available data in each analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
mg/L
  Baseline flare: hsCRP [N=107, 110] | 3.84 [3.26 to 4.53] | 6.38 [5.43 to 7.50]
  Baseline flare: SAA [N=95, 104] | 6.31 [4.95 to 8.04] | 15.85 [12.58 to 19.98]
  Last post-baseline flare: hsCRP [N= 22, 42] | 3.69 [2.44 to 5.60] | 4.32 [3.23 to 5.60]
  Last post-baseline flare: SAA, [N= 19, 39] | 6.74 [3.56 to 12.78] | 11.04 [7.17 to 17.02]

22. Secondary Outcome: Patient's Assessment of Gout Pain Intensity in the Most Affected Joint
Description: Participant scored their current pain intensity in the most affected joint of the gout flare on a 5-point Likert Scale (none, mild, moderate, severe, extreme).
Time Frame: 72 hours post-dose and 24 weeks post-dose
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
percentage of participants
  72 hours - None [N=108, 111] | 30.6 | 18.0
  72 hours - Mild [N=108, 111] | 48.1 | 45.0
  72 hours - Moderate [N=108, 111] | 20.4 | 27.0
  72 hours - Severe [N=108, 111] | 0.9 | 8.1
  72 hours - Extreme [N=108, 111] | 0.0 | 1.8
  24 weeks - None [N=79, 70] | 72.2 | 67.1
  24 weeks - Mild [N=79, 70] | 19.0 | 25.7
  24 weeks - Moderate [N=79, 70] | 6.3 | 7.1
  24 weeks - Severe [N=79, 70] | 2.5 | 0.0
  24 weeks - Extreme [N=79, 70] | 0.0 | 0.0

23. Secondary Outcome: Percentage of Patients With Maximum Severity of New Gout Flares as Severe or Extreme
Description: For each new flare, participants scored the maximum amount of acute gout pain in the most affected joint since the onset of the new flare and the time they were re-dosed on a 5 point Likert scale as None, Mild, Moderate, Severe or Extreme. The percentage of participants with a maximum new flare severity of severe or extreme is reported for the first post-baseline flare that occurred during the 12-week core study and for the last post-baseline flare that occurred up until the end of the first extension period.
Time Frame: From the onset of a new flare until re-dosing. First post-baseline new flare during 12 week core study and the last post-baseline flare that occurred up until the end of the first extension study (24 weeks).
Population: The number of participants analyzed (indicated by 'N') for the first new post-baseline flare includes patients who were re-treated for a new flare during the 12-week core study. For the last post-baseline flare the population analyzed includes patients re-treated for at least one new flare during the first 24 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 25 | 46
Percentage of participants
  First post-baseline flare [N= 12, 37] | 66.7 | 78.4
  Last post-baseline flare [N= 25, 46] | 64.0 | 78.3

24. Secondary Outcome: Time to First New Flare: Survival Analysis by Treatment Over 72 Weeks
Description: Kaplan-Meier estimates of time to first new flare and confidence intervals were determined. For patients with event, time to event = (date of event - date of first dose of study drug + 1).
  Patients met definition of new flare if they had:
  * Flare in joint, not a previously affected joint (at baseline or during study)
  * Flare in joint previously affected (at baseline or during study) after previous flare in joint has resolved completely.
  Patients did not meet criterion of having new gout flare if:
  • Increasing/renewed gout pain in an affected joint before flare has resolved completely.
Time Frame: From randomization to the end of the second extension period (72 weeks).
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
days | 254.0 [209.0 to 284.0] | 146.0 [94.0 to 202.0]

25. Secondary Outcome: Flare Rate Per Year
Description: Flare rate was calculated as the number of new flares over the period of observation in years. Flare rate was calculated using only those new flares before switching to canakinumab.
  Participants met the definition of new flare if they had:
  * Flare in joint, not a previously affected joint (at baseline or during study)
  * Flare in joint previously affected (at baseline or during study) after previous flare in joint has resolved completely.
  Participants did not meet criterion of having new gout flare if:
  • Increasing/renewed gout pain in an affected joint before the flare has resolved completely.
  Flare rates were estimated from a negative binomial model with body mass index at baseline as a covariate.
Time Frame: From randomization to the end of the second extension period (72 weeks).
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: flares per patient per year
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 112 | 114
flares per patient per year | 1.18 [0.96 to 1.45] | 2.02 [1.65 to 2.47]

26. Secondary Outcome: Patient's Assessment of Gout Pain Intensity for Participants Re-treated or Switched to Canakinumab
Description: Participants scored their current pain intensity in the most affected joint of the gout flare on a 5-point Likert Scale (none, mild, moderate, severe or extreme).
  Data are reported for the last post-baseline flare for participants who were randomized to and re-treated with canakinumab, and for the first post-baseline flare treated with canakinumab for participants randomized to triamcinolone acetonide and who were switched to canakinumab in extension study 2.
Time Frame: 72 hours post-dose and 7 days post dose for the last post-baseline flare for the canakinumab re-treated arm and for the first post-baseline flare treated with canakinumab in the triamcinolone acetonide arm during the overall 72 weeks.
Population: Modified Analysis Set (MAS) consisting of all FAS patients who were either re-treated or switched to canakinumab during the 72 weeks. At each timepoint only patients with a value at both baseline flare and the new flare are included.
Measure: Number; unit: percentage of participants
Groups:
- Re-treated With Canakinumab 150 mg: Participants who received canakinumab 150 mg in the core study and who were re-treated with canakinumab 150 mg for new flares during the overall 72 weeks. Data are reported for the last post-baseline flare for participants in this arm.
- Triam Switched to Canakinumab: Participants who received triamcinolone acetonide (triam) 40 mg in the core study and who were switched to canakinumab 150 mg for treatment of new flares in extension study 2. Data are reported for the first post-baseline flare treated with canakinumab.
Arm/Group | Re-treated With Canakinumab 150 mg | Triam Switched to Canakinumab
Number analyzed (Participants) | 62 | 41
percentage of participants
  72 hours - None [N=59, 40] | 30.5 | 25.0
  72 hours - Mild [N=59, 40] | 44.1 | 62.5
  72 hours - Moderate [N=59, 40] | 22.0 | 12.5
  72 hours - Severe [N=59, 40] | 3.4 | 0.0
  72 hours - Extreme [N=59, 40] | 0.0 | 0.0
  7 days - None [N=57, 37] | 64.9 | 59.5
  7 days - Mild [N=57, 37] | 21.1 | 35.1
  7 days - Moderate [N=57, 37] | 10.5 | 5.4
  7 days - Severe [N=57, 37] | 3.5 | 0.0
  7 days - Extreme [N=57, 37] | 0.0 | 0.0

27. Secondary Outcome: Patient's Global Assessment of Response to Treatment for Participants Re-treated or Switched to Canakinumab
Description: Participants made a global assessment of response to treatment using a 5-point Likert scale: Excellent, good, acceptable, slight or poor. Data are reported for the last post-baseline flare for participants who were randomized to and re-treated with canakinumab, and for the first post-baseline flare treated with canakinumab for participants randomized to triamcinolone acetonide and who were switched to canakinumab in extension study 2.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Re-treated With Canakinumab 150 mg | Triam Switched to Canakinumab
Number analyzed (Participants) | 62 | 41
percentage of participants
  72 hours - Excellent [N=58, 38] | 41.4 | 36.8
  72 hours - Good [N=58, 38] | 32.8 | 39.5
  72 hours - Acceptable [N=58, 38] | 12.1 | 21.1
  72 hours - Slight [N=58, 38] | 13.8 | 2.6
  72 hours - Poor [N=58, 38] | 0.0 | 0.0
  7 days - Excellent [N=56, 39] | 51.8 | 51.3
  7 days - Good [N=56, 39] | 26.8 | 33.3
  7 days - Acceptable [N=56, 39] | 10.7 | 7.7
  7 days - Slight [N=56, 39] | 7.1 | 7.7
  7 days - Poor [N=56, 39] | 3.6 | 0.0

28. Secondary Outcome: Physician's Global Assessment of Response to Treatment for Participants Re-treated or Switched to Canakinumab
Description: The study physician made a global assessment of the patient's response to treatment using a 5-point Likert scale: very good, good, fair, poor or very poor.
  The physician completed the physician's global assessment of response to treatment without viewing any of the patient's assessments.
  Data are reported for the last post-baseline flare for participants who were randomized to and re-treated with canakinumab, and for the first post-baseline flare treated with canakinumab for participants randomized to triamcinolone acetonide and who were switched to canakinumab in extension study 2.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Re-treated With Canakinumab 150 mg | Triam Switched to Canakinumab
Number analyzed (Participants) | 62 | 41
percentage of participants
  72 hours - Very good [N=56, 38] | 39.3 | 42.1
  72 hours - Good [N=56, 38] | 39.3 | 39.5
  72 hours - Fair [N=56, 38] | 16.1 | 18.4
  72 hours - Poor [N=56, 38] | 5.4 | 0.0
  72 hours - Very poor [N=56, 38] | 0.0 | 0.0
  7 days - Very good [N=58, 39] | 56.9 | 59.0
  7 days - Good [N=58, 39] | 25.9 | 38.5
  7 days - Fair [N=58, 39] | 15.5 | 2.6
  7 days - Poor [N=58, 39] | 1.7 | 0.0
  7 days - Very poor [N=58, 39] | 0.0 | 0.0

29. Secondary Outcome: Physician's Assessment of Joint Tenderness for Participants Re-treated or Switched to Canakinumab
Description: The study physician assessed the most affected joint for tenderness on the following 4-point scale:
  * no pain;
  * participant states that "there is pain;
  * participant states "there is pain and winces";
  * participant states "there is pain, winces and withdraws" on palpation or passive movement of the affected study joint.
  Data are reported for the last post-baseline flare for participants who were randomized to and re-treated with canakinumab, and for the first post-baseline flare treated with canakinumab for participants randomized to triamcinolone acetonide and who were switched to canakinumab in extension study 2.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Re-treated With Canakinumab 150 mg | Triam Switched to Canakinumab
Number analyzed (Participants) | 62 | 41
percentage of participants
  72 hours - No pain [N=56, 38] | 51.8 | 42.1
  72 hours - Pain [N=56, 38] | 37.5 | 50.0
  72 hours - Pain and winces [N=56, 38] | 5.4 | 5.3
  72 hours - Pain, winces and withdraws [N=56, 38] | 5.4 | 2.6
  7 days - No pain [N=58, 39] | 74.1 | 79.5
  7 days - Pain [N=58, 39] | 22.4 | 20.5
  7 days - Pain and winces [N=58, 39] | 3.4 | 0.0
  7 days - Pain, winces and withdraws [N=58, 39] | 0.0 | 0.0

30. Secondary Outcome: Physician's Assessment of Joint Swelling for Participants Re-treated or Switched to Canakinumab
Description: The study physician assessed the most affected joint for swelling on the following 4-point scale:
  * no swelling;
  * palpable;
  * visible;
  * bulging beyond the joint margins.
  Data are reported for the last post-baseline flare for participants who were randomized to and re-treated with canakinumab, and for the first post-baseline flare treated with canakinumab for participants randomized to triamcinolone acetonide and who were switched to canakinumab in extension study 2.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Re-treated With Canakinumab 150 mg | Triam Switched to Canakinumab
Number analyzed (Participants) | 62 | 41
percentage of participants
  72 hours - No swelling [N=56, 38] | 55.4 | 47.4
  72 hours - Palpable [N=56, 38] | 26.8 | 34.2
  72 hours - Visible [N=56, 38] | 12.5 | 15.8
  72 hours - Bulging beyond joint margins [N=56, 38] | 5.4 | 2.6
  7 days - No swelling [N=58, 39] | 70.7 | 79.5
  7 days - Palpable [N=58, 39] | 17.2 | 17.9
  7 days - Visible [N=58, 39] | 10.3 | 2.6
  7 days - Bulging beyond joint margins [N=58, 39] | 1.7 | 0.0

31. Secondary Outcome: Physician's Assessment of Erythema for Participants Re-treated or Switched to Canakinumab
Description: The study physician assessed the most affected joint for erythema (redness of the skin) as either present, absent or not assessable.
  Data are reported for the last post-baseline flare for participants who were randomized to and re-treated with canakinumab, and for the first post-baseline flare treated with canakinumab for participants randomized to triamcinolone acetonide and who were switched to canakinumab in extension study 2.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Re-treated With Canakinumab 150 mg | Triam Switched to Canakinumab
Number analyzed (Participants) | 62 | 41
percentage of participants
  72 hours - Absent [N=56, 38] | 73.2 | 92.1
  72 hours - Present [N=56, 38] | 26.8 | 7.9
  7 days - Absent [N=58, 39] | 84.5 | 94.9
  7 days - Present [N=58, 39] | 15.5 | 5.1

32. Secondary Outcome: High-sensitivity C-reactive Protein (hsCRP) Levels for Participants Re-treated With or Switched to Canakinumab
Description: High sensitivity C-reactive protein (hsCRP) levels in blood serum were measured by a central laboratory in order to identify the presence of inflammation, to determine its severity, and to monitor the response to treatment.
  Data are reported for the last post-baseline flare for participants who were randomized to and re-treated with canakinumab, and for the first post-baseline flare treated with canakinumab for participants randomized to triamcinolone acetonide and who were switched to canakinumab in extension study 2.
Time Frame: 24 hours, 72 hours, 7 days, 4, 8 and 12 weeks post-dose for the last post-baseline flare for the canakinumab re-treated arm and for the first post-baseline flare treated with canakinumab in the triamcinolone acetonide arm during the overall 72 weeks.
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Re-treated With Canakinumab 150 mg: Participants who received canakinumab 150 mg in the Ccre study and who were re-treated with canakinumab 150 mg for new flares during the overall 72 weeks. Data are reported for the last post-baseline flare for participants in this arm.
Arm/Group | Re-treated With Canakinumab 150 mg | Triam Switched to Canakinumab
Number analyzed (Participants) | 62 | 41
mg/L
  24-hours post-dose [N=48, 36] | 30.1 (64.11) | 39.4 (41.10)
  72-hours post-dose [N=56, 38] | 10.4 (31.11) | 12.6 (15.80)
  7 days post-dose [N=55, 40] | 2.8 (4.97) | 3.5 (5.00)
  4 weeks post-dose [N=46, 37] | 1.6 (2.30) | 2.2 (3.54)
  8 weeks post-dose [N=37, 35] | 2.1 (4.41) | 2.4 (4.62)
  12 weeks post-dose [N=38, 31] | 1.3 (0.79) | 2.9 (4.90)

33. Secondary Outcome: Serum Amyloid A Protein (SAA) Levels for Participants Re-treated With or Switched to Canakinumab
Description: Serum Amyloid A Protein (SAA) levels in blood serum were measured by a central laboratory in order to identify the presence of inflammation, to determine its severity, and to monitor the response to treatment.
  Data are reported for the last post-baseline flare for participants who were randomized to and re-treated with canakinumab, and for the first post-baseline flare treated with canakinumab for participants randomized to triamcinolone acetonide and who were switched to canakinumab in extension study 2.
Time Frame: as for outcome 32
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Re-treated With Canakinumab 150 mg | Triam Switched to Canakinumab
Number analyzed (Participants) | 62 | 41
mg/L
  24-hours post-dose [N=47, 36] | 129.0 (324.45) | 145.9 (257.44)
  72-hours post-dose [N=54, 37] | 45.6 (163.45) | 45.4 (97.00)
  7 days post-dose [N=56, 39] | 5.7 (8.90) | 5.9 (8.34)
  4 weeks post-dose [N=47, 37] | 3.4 (3.67) | 5.0 (7.02)
  8 weeks post-dose [N=38, 35] | 3.5 (4.24) | 5.3 (13.41)
  12 weeks post-dose [N=38, 29] | 3.4 (2.37) | 4.8 (5.94)

ADVERSE EVENTS:
Arm/Group | All Canakinumab | Canakinumab: Before Retreatment | Canakinumab: After Retreatment | All Triamcinolone Acetonide | Triam: Before Switch to Canakinumab | Triam: After Switch to Canakinumab
Serious Adverse Events (participants affected / at risk) | 12/112 | 1/62 | 5/62 | 4/114 | 0/41 | 3/41
Other Adverse Events (participants affected / at risk) | 42/112 | 15/62 | 19/62 | 36/114 | 15/41 | 8/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Canakinumab (N=112) | Canakinumab: Before Retreatment (N=62) | Canakinumab: After Retreatment (N=62) | All Triamcinolone Acetonide (N=114) | Triam: Before Switch to Canakinumab (N=41) | Triam: After Switch to Canakinumab (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Canakinumab (N=112) | Canakinumab: Before Retreatment (N=62) | Canakinumab: After Retreatment (N=62) | All Triamcinolone Acetonide (N=114) | Triam: Before Switch to Canakinumab (N=41) | Triam: After Switch to Canakinumab (N=41)
Nausea (Gastrointestinal disorders) | 3 | 2 | 1 | 3 | 1 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 5 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 9 | 4 | 7 | 3 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 3 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 5 | 10 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 2 | 6 | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 7 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 6 | 4 | 1
Headache (Nervous system disorders) | 5 | 3 | 2 | 6 | 2 | 1
Hypertension (Vascular disorders) | 14 | 3 | 7 | 7 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.